CLINICAL TRIAL: NCT02417571
Title: Effect of Ambulatory BP Monitoring on the CliniCal coUrse and RenAl ouTcomE of Chronic Kidney Disease
Brief Title: Effect of Ambulatory BP Monitoring on the CliniCal coUrse and RenAl ouTcomE of CKD
Acronym: ACCURATE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Kangbuk Samsung Hospital (Other); Severance Hospital (Other); Eulji General Hospital (Other)
Responsible Party: Principal Investigator, Kook-Hwan Oh, Associate professor, Division of Nephrology, Department of Internal Medicine, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BR-ABPM
Record Dates: First submitted 2015-04-11; First posted 2015-04-15 (Estimated); Last update posted 2019-06-05 (Actual); Status verified 2019-06

CONDITIONS: Chronic Kidney Diseases; Renal Insufficiency, Chronic; Albuminuria; Hypertension
Keywords: Chronic kidney disease; Blood pressure; ambulatory blood pressure; glomerular filtration rate
MeSH Terms: conditions — Renal Insufficiency, Chronic; Albuminuria; Hypertension | interventions — Blood Pressure Monitoring, Ambulatory

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ABPM group (Experimental): Ambulatory blood pressure monitoring (ABPM) performed at 3, 6 months after randomization; adjusting drugs/doses based on ABPM results.
  Target BP: daytime ABP < 135/85 mm Hg according to British NICE clinical guideline 127.
  Interventions: Device: Ambulatory blood pressure monitoring (ABPM)
- Office BP group (No Intervention): Conventional BP management using office BP according to KDIGO guideline on BP management.
  Target BP: <140/90 mm Hg.

INTERVENTIONS:
Device: Ambulatory blood pressure monitoring (ABPM) — 24-hour ambulatory BP monitoring using TM-2430 device (A&D Company, Tokyo, Japan)
  Arms: ABPM group

SUMMARY:
Control of blood pressure (BP) is the first thing to do in the management of chronic kidney disease (CKD). Although guidelines suggest the optimal blood pressure level, it is hard to assess BP correctly during the office visit. Often there is a discrepancy between office BP and out-of-office BP, including home BP and ambulatory BP. Recent study reported that as many as 34% of Korean CKD patients had masked hypertension, which means high BP by ambulatory BP monitoring but normal BP by conventional office BP measurement.

This study aims to evaluate the effect of ambulatory BP-guided BP management on the clinical outcome of CKD, compared to the conventional management using office BP.

DETAILED DESCRIPTION:
We hypothesized that management of blood pressure using ambulatory BP monitoring would obtain more optimal BP control and thereby would influence positively on renal progression and CV outcomes.

In detail, when the eligibility criteria is met, all the subjects will undergo both ambulatory BP and office BP measurement at baseline.

After randomization, ARB (fimasartan) will be administered to drug-naive subjects or will replace the other RAS blockers in subjects with current uses. Dosing of fimasartan will be adjusted or additional drugs of other classes will be added sequentially over 3 months (titration phase).

At 3 months, ABPM will be performed in ABPM group to evaluate the adequacy of blood pressure control and dosing will be adjusted according to the ABPM results (target BP: daytime BP < 135/85 mm Hg). This adjustment will be assessed at 6 months by ABPM once again.

For subjects in office BP group, conventional care will be provided according to current guidelines (target BP < 140/90 mm Hg).

At 18 months, ABPM will be performed in all the subjects and outcome measures will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Office BP > 130/80 mm Hg, irrespective of anti-hypertensive medication
* CKD stages 3-4 (or estimated GFR 15-59 ml/min per 1.73 m2)
* Random urine albumin-to-creatinine ratio > 300 mg/g or protein-to-creatinine ration > 300 mg/g or dipstick albumin > 1+, in case of estimated GFR 45-59 ml/min per 1.73 m2

Exclusion Criteria:

* Systolic BP > 180 mm Hg or diastolic BP > 110 mm Hg
* Malignant hypertension
* Resistant hypertension (using more than three kind of anti-hypertensive drugs other than diuretics)
* Uncontrolled DM (Hb A1c > 10.0% within 3 months of eligibility assessment)
* Use of immunosuppressive agents within 1 months or anticipated
* Atrial fibrillation or flutter
* Contraindication to renin-angiotensin system blockers (hypersensitivity, bilateral renal artery stenosis, single kidney, etc.)
* Pregnancy
* Kidney recipients
* Participating other clinical trials, except observational studies

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Estimated)
Dates: Start 2015-04 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
rate of estimated GFR decline | 18 months
  annual decline of eGFR over 18 months

SECONDARY OUTCOMES:
Renal events | 18 months
  dialysis, transplantation, doubling of serum creatinine or >50% decline of eGFR
Albuminuria | 18 months
  change of urine albumin-to-creatinine ratio
CV events | 18 months
  Cardiovascular deaths, nonfatal myocardial infarction, admission due to aggravation of CHF, or revascularization (CABG or PCI)
All-cause mortality | 18 months

CONTACTS AND LOCATIONS:
Locations (4):
- South Korea (4):
  - Eulji General Hospital, Seoul
  - Kangbuk Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Yonsei University Severance Hospital, Seoul

REFERENCES:
- [Background] Cha RH, Kim S, Ae Yoon S, Ryu DR, Eun Oh J, Han SY, Young Lee E, Ki Kim D, Kim YS. Association between blood pressure and target organ damage in patients with chronic kidney disease and hypertension: results of the APrODiTe study. Hypertens Res. 2014 Feb;37(2):172-8. doi: 10.1038/hr.2013.127. Epub 2013 Sep 19. PMID 24048482
- [Derived] Kim Y, Kim J, Kang E, Im DW, Kim T, Huh H, Kim YH, Lee H, Kim JH, Oh KH. The association of time-updated ambulatory blood pressure and renal progression in hypertensive patients with chronic kidney disease: post hoc analysis of ACCURATE study. J Hypertens. 2024 Mar 1;42(3):515-520. doi: 10.1097/HJH.0000000000003625. Epub 2023 Dec 6. PMID 38088422
- [Derived] Kim Y, Kim J, Lee SW, Sung S, Yoo TH, Lee KB, Hwang YH, Kim T, Kang SW, Kim YH, Oh KH. Effect of ambulatory blood pressure monitoring guided antihypertensive treatment on renal progression in patients with chronic kidney disease: a randomized comparative study. J Hypertens. 2021 Feb 1;39(2):325-332. doi: 10.1097/HJH.0000000000002624. PMID 33031169
- See also: 2012 KDIGO Clinical Practice Guideline for the Management of Blood Pressure in Chronic Kidney Disease — https://kdigo.org/guidelines/blood-pressure-in-ckd/
- See also: British NICE guideline 127: Hypertension: clinical management of primary hypertension in adults — http://www.nice.org.uk/guidance/CG127